CLINICAL TRIAL: NCT02245828
Title: A Randomized, Double-blind, Placebo-controlled First-in-human Study to Assess the Safety, Tolerability and Pharmacokinetics of Single and Multiple Ascending Doses of QCC374 in Healthy Subjects
Brief Title: A First in Human Study to Assess the Safety, Tolerability and Pharmacokinetics of Single and Multiple Ascending Doses of QCC374
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CQCC374X2101
Record Dates: First submitted 2014-08-28; First posted 2014-09-22 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-03

CONDITIONS: Healthy Subjects
Keywords: healthy subjects, inhaled
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo comparator
  Interventions: Drug: Placebo
- QCC374 (Experimental): Single and multiple ascending doses of QCC374
  Interventions: Drug: QCC374

INTERVENTIONS:
Drug: QCC374 — Single and multiple ascending doses of QCC374
  Arms: QCC374
Drug: Placebo — Placebo comparator
  Arms: Placebo

SUMMARY:
This is a double blind, randomized, placebo controlled, single and multiple ascending dose study in healthy subjects. Safety evaluation will include (serious) adverse events, vital signs, body weight and lung function tests. Blood samples for Pharmacokinetics will also be drawn at specified timepoints.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be obtained before any assessment is performed.
2. Healthy male and female subjects age 18 to 55 years of age included, and in good health as determined by past medical history, physical examination, vital signs, electrocardiogram, and laboratory tests at screening.
3. Weight of at least 50 kg and body mass index (BMI) within the range of 18 - 32 kg/m2. BMI = Body weight (kg) / [Height (m)]2.
4. Oxygen saturation (O2) at screening must be ≥ 95% on room air.
5. FEV1 ≥ 90% predicted.

Exclusion Criteria:

1. 1. A history of clinically significant ECG abnormalities and/or orthostatic vital signs at screening.
2. History of asthma or reactive airway diseases.
3. Smokers or anyone who smoked within 5 years of screening. Urine cotinine levels ≥ 500 ng/mL.
4. History of malignancy of any organ system other than localized basal cell carcinoma of the skin, treated or untreated within the past 5 years, regardless of whether there is evidence of local recurrence or metastases.
5. Women of child-bearing potential

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2014-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | 39 days
  Number of Participants with Adverse Events

SECONDARY OUTCOMES:
AUCinf | 39 days
  Area under the plasma concentration-time curve from time zero to infinity
AUClast | 39 days
  The area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration
AUCtau | 39 days
  The area under the plasma concentration-time curve from time zero to the end of the dosing interval tau
Cav | 39 days
  The average steady state plasma concentration during multiple dosing
Cmax | 39 days
  The observed maximum plasma concentration following drug administration
T1/2 | 39 days
  The terminal elimination half life
Tmax | 39 days
  The time to reach the maximum concentration after drug administration

CONTACTS AND LOCATIONS:
Locations (1):
- Novartis Investigative Site, Mid Glamorgan, Wales, United Kingdom